CLINICAL TRIAL: NCT00866177
Title: Phase II Trial of Hyd-sulfate AZD6244 [NSC 748727] in Patients With BRAF or NRAS Mutated Melanomas
Brief Title: MEK Inhibitor AZD6244 in Treating Patients With Stage III or Stage IV Melanoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2009-01164; NCI-2009-01164 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); MSKCC-09003; CDR0000637669; 09-003 (Other: Memorial Sloan-Kettering Cancer Center); 8252 (Other: CTEP); N01CM62206 (NIH); P30CA008748 (NIH)
Record Dates: First submitted 2009-03-19; First posted 2009-03-20 (Estimated); Results first posted 2015-08-11 (Estimated); Last update posted 2015-08-11 (Estimated); Status verified 2013-06

CONDITIONS: Recurrent Melanoma; Stage III Skin Melanoma; Stage IV Skin Melanoma
MeSH Terms: conditions — Melanoma | interventions — AZD 6244

ARMS (1):
- Arm I (Experimental): Patients receive oral MEK inhibitor AZD6244 twice daily on days 1-28. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Other: Laboratory Biomarker Analysis; Drug: Selumetinib

INTERVENTIONS:
Other: Laboratory Biomarker Analysis — Correlative studies
Drug: Selumetinib — Given orally
  Other Names: ARRY-142886; AZD6244; MEK Inhibitor AZD6244

SUMMARY:
This phase II trial is studying how well MEK inhibitor AZD6244 works in treating patients with stage III or stage IV melanoma. MEK inhibitor AZD6244 may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Determine the response in patients with V600E or V600K BRAF-mutated or NRAS-mutated stage III or stage IV melanoma with low or high phospho-pAKT expression treated with MEK inhibitor AZD6244.

SECONDARY OBJECTIVES:

I. Identify other genetic predictors of sensitivity to MEK inhibition.

OUTLINE: Patients are stratified according to pAKT expression (low vs high).

Patients receive oral MEK inhibitor AZD6244 twice daily on days 1-28. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.

Tumor tissue samples are collected for correlative laboratory studies. Samples are assessed for expression of pAKT, pPRAS40, and PTEN by IHC and mutations in BRAF, NRAS, KIT, and PIK3CAP by MALDI-TOF. PTEN is sequenced in tumors using whole genome amplification followed by high-throughput bidirectional dideoxynucleotide sequencing of PCR-amplified gene products.

After completion of study treatment, patients are followed for 4 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed melanoma

  * Stage IV or stage III disease not potentially curable with surgery
* Documented tumor progression
* Must have a V600E or V600K BRAF-mutated tumor, or a NRAS mutation at condons 12, 13, or 61
* Measurable disease, defined as ≥ 1 unidimensionally measurable lesion ≥ 20 mm by conventional techniques or ≥ 10 mm by spiral CT scan
* Must have tumor tissue (block or unstained slides) available for IHC studies
* No primary uveal or mucosal melanoma
* No active or untreated brain metastases

  * Treated brain metastases allowed provided they have been stable for ≥ 3 months
* ECOG performance status 0-1
* Life expectancy > 3 months
* WBC ≥ 3,000/mcL
* Absolute neutrophil count ≥ 1,500/mcL
* Platelet count ≥ 100,000/mcL
* Hemoglobin ≥ 9.0 g/dL (no requirement for transfusions within the past 2 weeks)
* Total bilirubin ≤ 1.5 times upper limit of normal (ULN)
* AST/ALT ≤ 2.5 times ULN
* Creatinine ≤ 1.5 mg/dL
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception during and for 16 weeks after completion of study treatment
* No refractory nausea and vomiting, chronic gastrointestinal disease (e.g., inflammatory bowel disease), or significant bowel resection that would preclude adequate absorption
* No concurrent uncontrolled illness, including, but not limited to, any of the following:

  * Ongoing or active infection or bleeding
  * Symptomatic congestive heart failure
  * Unstable angina pectoris
  * Cardiac arrhythmia
  * Psychiatric illness/social situation that would limit compliance with study requirements
* No history of allergic reactions attributed to compounds of similar chemical or biologic composition to MEK inhibitor AZD6244
* Any number of prior therapies allowed
* At least 4 weeks since prior radiotherapy or chemotherapy (6 weeks for nitrosoureas or mitomycin C) and recovered
* At least 4 months since prior anti-CTLA4 monoclonal antibody therapy
* At least 4 weeks since other prior systemic therapy
* No other concurrent investigational agents
* No concurrent antiretroviral therapy for HIV-positive patients
* No concurrent vitamin E supplementation or multivitamin supplements that provide a total daily dose in excess of 100% of the recommended daily dose of vitamin E
* No concurrent anticancer chemotherapy or other systemic drugs
* Concurrent palliative radiotherapy allowed

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 167 (Actual)
Dates: Start 2009-03; Primary Completion 2013-09 (Actual); Study Completion 2013-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Paul Chapman, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan-Kettering Cancer Center, New York, New York, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- AZD6244: Patients receive oral MEK inhibitor AZD6244 twice daily on days 1-28. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.
Period: Overall Study
Arm/Group | AZD6244
Started | 167
Completed | 15
Not Completed | 152
Not completed — Withdrawal by Subject | 1
Not completed — Not Treated | 151

BASELINE CHARACTERISTICS:
Arm/Group | AZD6244
Number analyzed (Participants) | 167
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 107
  >=65 years | 60
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 51
  Male | 116
Region of Enrollment [Number; unit: participants]
  United States | 167

OUTCOME MEASURES:

1. Primary Outcome: Anti-tumor Response Defined as Either a CR, PR, or SD as Defined by RECIST
Description: Anti-tumor response defined as either a Complete Response, Partial Response, or Stable Disease as defined by RECIST
Time Frame: Up to 4 weeks
Measure: Number; unit: participants
Arm/Group | AZD6244
Number analyzed (Participants) | 15
participants
  Partial Response | 1
  Stable Disease | 8
  Progression of Disease | 6

ADVERSE EVENTS:
Arm/Group | AZD6244
Serious Adverse Events (participants affected / at risk) | 6/15
Other Adverse Events (participants affected / at risk) | 14/15
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | AZD6244 (N=15)
Alanine aminotransferase increased (Investigations) | 2 (2)
Aspartate aminotransferase increased (Investigations) | 2 (2)
Alkaline phosphatase increased (Investigations) | 1 (2)
Blood Bilirubin increase (Investigations) | 1 (2)
Diarrhea (Gastrointestinal disorders) | 1 (1)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (3)
Fatigue (General disorders) | 1 (1)
Fever (General disorders) | 1 (2)
Heart failure (Cardiac disorders) | 1 (1)
Left ventricular systolic dysfunction (Cardiac disorders) | 2 (2)
Neoplasms benign, malignant and unspecified (incl cysts and polyps) - Other, specify (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2)
Chest pain (General disorders) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Rash, acne (Skin and subcutaneous tissue disorders) | 1 (1)
Right ventricular dysfunction (Cardiac disorders) | 1 (1)
Rigors/chills (General disorders) | 1 (1)
Thromboembolic event (Vascular disorders) | 1 (1)
Vascular disorder (Vascular disorders) | 2 (2)
Vomiting (Gastrointestinal disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | AZD6244 (N=15)
Alanine aminotransferase increased (Investigations) | 9 (14)
Alkaline phosphatase increased (Investigations) | 8 (24)
Aspartate aminotransferase increased (Investigations) | 10 (30)
Alopecia (Skin and subcutaneous tissue disorders) | 1 (1)
Anemia (Blood and lymphatic system disorders) | 8 (16)
Blood Bilirubin increased (Investigations) | 5 (10)
Cardiac disorder (Cardiac disorders) | 1 (1)
Chest wall pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Constipation (Gastrointestinal disorders) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 3 (3)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 4 (5)
Edema-Limbs (General disorders) | 2 (2)
Fatigue (General disorders) | 5 (6)
Fever (General disorders) | 1 (1)
Heart failure (Cardiac disorders) | 1 (1)
Hyperglycemia (Metabolism and nutrition disorders) | 6 (22)
Hyperkalemia (Metabolism and nutrition disorders) | 1 (1)
Hypoalbuminemia (Metabolism and nutrition disorders) | 2 (6)
Hypocalcemia (Metabolism and nutrition disorders) | 1 (2)
Hypokalemia (Metabolism and nutrition disorders) | 2 (2)
Hypomagnesemia (Metabolism and nutrition disorders) | 4 (10)
Hypophosphatemia (Metabolism and nutrition disorders) | 1 (2)
INR increase (Investigations) | 1 (3)
Left ventricular systolic dysfunction (Cardiac disorders) | 2 (2)
Lymphocyte count decrease (Investigations) | 3 (3)
Nausea (Gastrointestinal disorders) | 2 (2)
Neutrophil count decrease (Investigations) | 1 (1)
Platelet count decrease (Investigations) | 3 (10)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Rash acneiform (Skin and subcutaneous tissue disorders) | 10 (12)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 2 (2)
Right ventricular dysfunction (Cardiac disorders) | 1 (1)
Skin ulceration (Skin and subcutaneous tissue disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 2 (2)
White blood cell decrease (Investigations) | 4 (6)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less